CLINICAL TRIAL: NCT00094406
Title: Effects of Inhaled Carbon Monoxide on Pulmonary Inflammatory Responses Following Endotoxin Instillation
Brief Title: Carbon Monoxide to Prevent Lung Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 050012; 05-CC-0012
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-04-19

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Lung Permeability; Endotoxin Tolerance; Bronchoscopy; Carbon Monoxide Inhalation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Bronchoscopy; Bronchoalveolar Lavage; Endotoxins; Carbon Monoxide

INTERVENTIONS:
Procedure: Bronchoscopy
Procedure: Bronchoalveolar lavage
Drug: Endotoxin
Drug: Carbon Monoxide

SUMMARY:
This study will examine in healthy volunteers how breathing carbon monoxide (CO) affects lung inflammation. Severe lung inflammation sometimes develops in patients with pneumonia or patients who develop serious blood stream infections. Studies in the laboratory and in animals show that CO can decrease lung inflammation.

Healthy volunteers between 18 and 40 years of age who do not smoke, are not taking any medications, do not have asthma, are not allergic to sulfa- and penicillin-based drugs, and are not pregnant may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), and chest x-ray. Subjects are enrolled in either a pilot study or the main study.

Participants undergo bronchoscopy and bronchoalveolar lavage to study the effects of endotoxin (a component of bacteria that causes inflammation similar to that in patients with lung infections) on lung function. Before the procedure, a small plastic tube (catheter) is placed in a vein to collect blood samples and another is placed in an artery to check blood pressure. For the bronchoscopy, the mouth and nasal airways are numbed with lidocaine, and a bronchoscope (thin flexible tube) is passed through the nose into the airways of the lung. A small amount of salt water is squirted through the bronchoscope into one lung and then salt water containing endotoxin is squirted into the other lung.

Following the bronchoscopy, subjects are treated with either CO or room air (placebo) for 6 hours. (Subjects in the pilot study receive treatment for only 3 hours). The gas is delivered through a cushioned mask placed over the nose and mouth. The amount of exhaled CO is measured before, during, and after inhalation of the gas. For this measurement, subjects take a deep breath to fill up their lungs and slowly exhale into a mouthpiece connected to a measuring device until they feel their lungs are empty.

After the CO treatment, a second bronchoscopy is done to examine how the lung responded to the CO or room air. This is studied in two ways. To sample the air, a large needle is used to withdraw air through the bronchoscope over about 3 seconds. Then the areas of the lung that were squirted with salt water alone and with endotoxin and salt water and are rinsed (lavage) and cells and secretions are collected.

...

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a major cause of morbidity and mortality. Of the many potential predisposing factors, sepsis and pneumonia represent the two main causes of ARDS. In spite of an increase in survival in recent years mortality in patients with ARDS is still estimated around 30 to 40%. In this context, development of effective preventive strategies in patients at high risk of development of ARDS is of paramount importance. Unfortunately, the results of studies evaluating prophylactic regimens for ARDS have been mostly disappointing.

The gaseous molecule carbon monoxide (CO) has been traditionally viewed as a toxic metabolic and industrial waste. However, recent studies have demonstrated an important physiologic role of CO in many biological systems. Specifically, strong anti-inflammatory, anti-oxidant and anti-thrombotic effects of CO gas administration and heme oxygenase activation (the enzyme that generates endogenous CO gas) have been demonstrated in several animal models.

Previous studies conducted in our department have demonstrated that bronchoscopic instillation of endotoxin (LPS) in healthy volunteers elicits a compartmentalized pulmonary inflammatory response, serving as an excellent model to evaluate interventions directed towards suppression of lung inflammation at its earliest stages.

In the current single blinded, randomized, placebo controlled study, we are planning to evaluate the effects of inhaled carbon monoxide on local pulmonary inflammatory responses following endotoxin administration. Healthy subjects will undergo local endotoxin instillation, breathe CO or room air through a mask for 6 hours, and then a repeat bronchoscopy with lavage will be done at 6 hours to assess the ability of CO to suppress local inflammation in the lung.

ELIGIBILITY:
* INCLUSION CRITERIA:

All volunteer subjects, employees and non-employees, must 18 to 40 years of age and must be able to provide informed, written consent for participation in this study. We will not directly advertise the study to employees to avoid the potential for coercion. Eligibility in the study is determined prior to enrollment on the basis of the following inclusion and exclusion criteria.

Normal screening examination including:

1. medical history and physical examination, nonsmoker, no concurrent medications including aspirin or nonsteroidal anti-inflammatory drugs, no active medical problems
2. complete blood count with differential and platelet counts
3. serum chemistries including creatinine, blood urea nitrogen, glucose, liver enzymes and function tests, electrolytes, prothrombin time, partial thromboplastin time, carboxyhemoglobin measured by venous co-oxymetry.
4. urinalysis
5. female subjects must have negative urine pregnancy test within one week of participation (this will be repeated immediately prior to beginning the screening procedures due to radiation exposure from the chest x-ray)
6. electrocardiogram
7. chest radiograph

Sexually active females not using contraceptive methods will be instructed to abstain from sexual activity or use barrier contraception methods from the time of last negative pregnancy test to 24 hours after completion of the study.

EXCLUSION CRITERIA:

1. active tobacco use
2. baseline caroxyhemoglobin greater than 2%
3. pregnancy
4. lactation
5. medical history of recent clinically significant asthma allergy to both sulfa- and penicillin-based drugs
6. Allergy to both sulfa- and penicillin-based drugs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-10-13; Primary Completion 2010-03-11 (Actual); Study Completion 2010-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Suffredini, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hudson LD, Milberg JA, Anardi D, Maunder RJ. Clinical risks for development of the acute respiratory distress syndrome. Am J Respir Crit Care Med. 1995 Feb;151(2 Pt 1):293-301. doi: 10.1164/ajrccm.151.2.7842182.
- [Background] Baumann WR, Jung RC, Koss M, Boylen CT, Navarro L, Sharma OP. Incidence and mortality of adult respiratory distress syndrome: a prospective analysis from a large metropolitan hospital. Crit Care Med. 1986 Jan;14(1):1-4. doi: 10.1097/00003246-198601000-00001. PMID 3484443
- [Background] Milberg JA, Davis DR, Steinberg KP, Hudson LD. Improved survival of patients with acute respiratory distress syndrome (ARDS): 1983-1993. JAMA. 1995 Jan 25;273(4):306-9. PMID 7815658
- [Derived] Zhang T, Zhang G, Chen X, Chen Z, Tan AY, Lin A, Zhang C, Torres LK, Bajrami S, Zhang T, Zhang G, Xiang JZ, Hissong EM, Chen YT, Li Y, Du YN. Low-dose carbon monoxide suppresses metastatic progression of disseminated cancer cells. Cancer Lett. 2022 Oct 10;546:215831. doi: 10.1016/j.canlet.2022.215831. Epub 2022 Jul 19. PMID 35868533